CLINICAL TRIAL: NCT05280197
Title: Benefit of Intraoperative TAP Blocks for Kidney Transplantation- a Randomized, Placebo Controlled Trial
Brief Title: Does an Abdominal Wall Nerve Block During Surgery Help Reduce Pain From Kidney Transplantation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Mohamed Eltemamy, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 21-748
Record Dates: First submitted 2022-01-11; First posted 2022-03-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplant; Renal Transplant; Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The surgeon performing the TAP block will be unblinded. The participant, investigators, and outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- liposomal bupivacaine plus free bupivacaine (Experimental)
  Interventions: Procedure: TAP block; Drug: liposomal bupivacaine plus free bupivacaine
- normal saline (Placebo Comparator)
  Interventions: Procedure: TAP block; Drug: normal saline

INTERVENTIONS:
Procedure: TAP block — Transversus abdominis plane (TAP) nerve block with liposomal bupivacaine plus free bupivacaine
  Arms: liposomal bupivacaine plus free bupivacaine
Procedure: TAP block — Transversus abdominis plane (TAP) nerve block with normal saline
  Arms: normal saline
Drug: liposomal bupivacaine plus free bupivacaine — TAP block using liposomal bupivacaine plus free bupivacaine
  Arms: liposomal bupivacaine plus free bupivacaine
Drug: normal saline — TAP block using normal saline
  Arms: normal saline

SUMMARY:
This is a randomized, placebo controlled, double blind study to determine the effectiveness of a Transversus Abdominis Plane (TAP) block for reducing postoperative pain and opioid use in kidney transplant recipients.

DETAILED DESCRIPTION:
The management of post-operative analgesia in kidney transplant recipients is complex secondary to labile fluid shifts and limitations in the use of NSAIDs secondary to their potential nephrotoxicity. A majority of transplant centers rely on the use of intravenous patient-controlled opioid analgesia as the predominant method of post-operative pain control, however this practice is at odds with the worldwide initiatives to reduce post-operative opioid use and dependence.

This study is a single center prospective randomized double blinded study which will compare the post-operative benefits of TAP block with liposomal bupivacaine plus free bupivacaine versus placebo (normal saline) TAP block in participants receiving both the ARS and the Gibson incisions for kidney transplantation . Approximately 200 participants will be enrolled at the Cleveland Clinic.

The operative approach (i.e. Gibson or ARS) is at the discretion of the operating surgeon and will proceed in the standard fashion. At the completion of the dissection of the external iliac vessels and prior to bringing the transplant kidney into the field, an intraoperative TAP block will be performed by inserting a 22 gauge spinal needle from inside the abdomen into the transversus abdominus plane of the abdominal wall at the lateral superior and inferior border of the surgical dissection and injecting the pre-determined analgesic or placebo.

The remainder of the procedure, including the vascular and urinary anastomosis, will proceed identically between the two groups. All participants will receive the same post-operative abdominal surgical dressing.

Post-operative pain control will follow standard clinical guidelines. All participants will be prescribed on-demand oral Oxycodone 5 or 10 mg tablets plus IV Morphine or IV Dilaudid if needed for severe breakthrough pain. On discharge, all participants will receive ten 5 or 10 mg Oxycodone tablets.

ELIGIBILITY:
Inclusion Criteria:

- Recipients of a single, living or deceased renal transplantation

Exclusion Criteria:

* Previous renal transplantation on the same side of the body
* Requiring a native or graft nephrectomy or other additional procedures
* Urine diversion or augmentation
* Bowel diversion
* Recipients of an enbloc pediatric kidney
* Recipients of a dual kidney transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Number of morphine milligram equivalents (MME) used in the post-operative period | Daily from the day after transplant (Post operative day 1) until day of discharge or 7 days, whichever comes first: Post-op Day 1
Number of morphine milligram equivalents (MME) used in the post-operative period | Daily from the day after transplant (Post operative day 1) until day of discharge or 7 days, whichever comes first: Post-op Day 2
Number of morphine milligram equivalents (MME) used in the post-operative period | Daily from the day after transplant (Post operative day 1) until day of discharge or 7 days, whichever comes first: Post-op Day 3
Number of morphine milligram equivalents (MME) used in the post-operative period | Daily from the day after transplant (Post operative day 1) until day of discharge or 7 days, whichever comes first: Post-op Day 4
Number of morphine milligram equivalents (MME) used in the post-operative period | Daily from the day after transplant (Post operative day 1) until day of discharge or 7 days, whichever comes first: Post-op Day 5
Number of morphine milligram equivalents (MME) used in the post-operative period | Daily from the day after transplant (Post operative day 1) until day of discharge or 7 days, whichever comes first: Post-op Day 6
Number of morphine milligram equivalents (MME) used in the post-operative period | Daily from the day after transplant (Post operative day 1) until day of discharge or 7 days, whichever comes first: Post-op Day 7
Number of morphine milligram equivalents (MME) used in the post-operative period | Twice weekly for 3 weeks, starting starting 1 week after transplant: Post-Op Week 2-1
Number of morphine milligram equivalents (MME) used in the post-operative period | Twice weekly for 3 weeks, starting starting 1 week after transplant: Post-Op Week 2-2
Number of morphine milligram equivalents (MME) used in the post-operative period | Twice weekly for 3 weeks, starting starting 1 week after transplant: Post-Op Week 3-1
Number of morphine milligram equivalents (MME) used in the post-operative period | Twice weekly for 3 weeks, starting starting 1 week after transplant: Post-Op Week 3-2
Number of morphine milligram equivalents (MME) used in the post-operative period | Twice weekly for 3 weeks, starting starting 1 week after transplant: Post-Op Week 4-1
Number of morphine milligram equivalents (MME) used in the post-operative period | Twice weekly for 3 weeks, starting starting 1 week after transplant: Post-Op Week 4-2
Number of morphine milligram equivalents (MME) used in the post-operative period | Every 2 weeks for 2 months, starting 1 month after the transplant date: Month 2, Week 2
Number of morphine milligram equivalents (MME) used in the post-operative period | Every 2 weeks for 2 months, starting 1 month after the transplant date: Month 2, Week 4
Number of morphine milligram equivalents (MME) used in the post-operative period | Every 2 weeks for 2 months, starting 1 month after the transplant date: Month 3, Week 2
Number of morphine milligram equivalents (MME) used in the post-operative period | Every 2 weeks for 2 months, starting 1 month after the transplant date: Month 3, Week 4
Number of morphine milligram equivalents (MME) used in the post-operative period | At 6 months after the transplant date
Number of morphine milligram equivalents (MME) used in the post-operative period | At 12 months after the transplant date

SECONDARY OUTCOMES:
Level of postoperative pain using using an adapted version of the brief pain inventory (BPI) which uses a 10-point numeric scale from 0-10. | Daily from the day after transplant (Post operative day 1) until day of discharge or 7 days, whichever comes first, then weekly for 3 weeks, then every 2 weeks for 2 months, then at 6 months and 12 month post surgical date
  The adapted brief pain inventory (BPI) uses a 10-point numeric scale, from 0-10. 0 indicates no pain and is the best outcome, 10 indicates the worst pain and is the worst outcome.

OTHER OUTCOMES:
Incidence of post-operative nausea and vomiting | Daily from the day after transplant (Post operative day 1) until day of discharge or 7 days, whichever comes first, then weekly for 3 weeks, then every 2 weeks for 2 months, then at 6 months and 12 month post surgical date
Incidence of post-operative ileus | Daily from the day after transplant (Post operative day 1) until day of discharge or 7 days, whichever comes first, then weekly for 3 weeks, then every 2 weeks for 2 months, then at 6 months and 12 month post surgical date
Length of post-operative hospital stay | Daily from the day after transplant (Post operative day 1) until day of discharge or 30 days, whichever comes first,

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Eltemamy, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams M, Milner QJ. Postoperative analgesia following renal transplantation - current practice in the UK. Anaesthesia. 2003 Jul;58(7):712-3. doi: 10.1046/j.1365-2044.2003.32661.x. No abstract available. PMID 12790818
- [Background] Singh PM, Borle A, Makkar JK, Trisha A, Sinha A. Evaluation of transversus abdominis plane block for renal transplant recipients - A meta-analysis and trial sequential analysis of published studies. Saudi J Anaesth. 2018 Apr-Jun;12(2):261-271. doi: 10.4103/sja.SJA_598_17. PMID 29628838
- [Background] Phillips SH, Hill SK, Lipscomb LD, Africa JB. First experience: Open small incision rectus sheath approach renal transplant: A case series. Int J Surg. 2017 Mar;39:114-118. doi: 10.1016/j.ijsu.2017.01.076. Epub 2017 Jan 18. PMID 28110032